CLINICAL TRIAL: NCT03674866
Title: A Canadian Multi-centre, Retrospective, Non-interventional Study of the Effectiveness of Tresiba® (Insulin Degludec) After Switching Basal Insulin in a Population With Type 1 or Type 2 Diabetes Mellitus CAN-TREAT (CANadian TREsiba AudiT)
Brief Title: A Canadian Study of the Effectiveness of Tresiba® (Insulin Degludec) After Switching Basal Insulin in a Population With Type 1 or Type 2 Diabetes Mellitus
Acronym: CAN-TREAT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4396; U1111-1203-7872 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes: Patients with type 1 diabetes and type 2 diabetes who received at least one prescription of insulin degludec (Tresiba®).
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec — Participants are treated with Tresiba® (insulin degludec) under conditions of routine care.

SUMMARY:
The purpose of this study is to collect historical data in real life conditions in a large group of people who have type 1 or type 2 diabetes and were treated with Tresiba® (insulin degludec) for at least 6 months. Data will be collected beginning 6 months before the participant started Tresiba® up to around 6 months after the participant started taking insulin degludec.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained before any study-related activities. Study-related activities are any data collection from the medical records of the patient
* Male or female age greater than or equal to 18 years at the time of insulin degludec initiation
* Type 1 diabetes mellitus or insulin-treated type 2 diabetes mellitus patients
* Switched to insulin degludec (± prandial insulin) after any basal insulin (± prandial insulin). Switch must have occurred at least 6 months prior to data collection and the patient may or may not be treated with insulin degludec at the time of patient selection
* Previously treated with any basal insulin (± prandial insulin) for at least 6 months prior to switching to insulin degludec
* At least one documented medical visit in the first 6 months (closest value in 3 to 9 months window) after insulin degludec initiation
* Minimum available data at the time of insulin degludec initiation: age, type of diabetes, HbA1c, duration of diabetes, duration and type of insulin treatment, medical follow-up at the study site for at least 1 year, and an estimated glomerular filtration rate (eGFR) value in the last 12 ±6 months (full data period)

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having signed the Informed Consent in this study
* Patients treated by continuous subcutaneous insulin infusion or premix insulin in the 6 months prior to receiving Tresiba

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes mellitus whose basal insulin was switched to insulin degludec
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  measured in % point

SECONDARY OUTCOMES:
Change in percentage of patients with HbA1c below 7% | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  percentage of patients
Change in percentage of patients with HbA1c below 7.5% | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  percentage of patients
Change in percentage of patients with HbA1c below 8.0% | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  percentage of patients
Change in the mean Fasting Plasma Glucose (FPG) | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  measured in mmol/L
Insulin degludec dose | At switch to insulin degludec (week 0)
  measured in units/day
Insulin degludec dose | 6 months after switch to insulin degludec
  measured in units/day
Change in the mean daily insulin doses (total, basal, prandial) | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  measured in units/day
Change in the number of concomitant non-insulin glucose-lowering drug classes | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  number of concomitant non-insulin glucose-lowering drug classes
Change in body weight | Baseline (up to 3 months prior to switch), 6 months after switch to insulin degludec
  measured in kg
Change in the percentage of patients with at least one hypoglycaemic episode (overall, nonsevere,non-severe) | Before change to insulin degludec (-6 to 0 months)
  percentage of patients
Change in the percentage of patients with at least one hypoglycaemic episode (overall, nonsevere,non-severe) | After change to insulin degludec (0 to 6 months)
  percentage of patients
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) | Before change to insulin degludec (-6 to 0 months)
  rates of hypoglycaemic episodes
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) | After change to insulin degludec (0 to 6 months)
  rates of hypoglycaemic episodes
Percentage of patients continuing insulin degludec | After change to insulin degludec (0 to 6 months)
  percentage of patients
Reason(s) for starting insulin degludec | At time of switch to insulin degludec (week 0)
  Reasons for starting insulin degludec (if available) will be classified as: Not at glycaemic target, Hypoglycaemia (severe / non-severe / nocturnal), Hypoglycaemia unawareness, Multiple risk factors for hypoglycaemia (elderly, intensive exercise, Chronic Kidney Disease, other), Basal insulin dose more than 80 units/day, Twice daily basal insulin dosing, Fasting blood glucose variability, Need for flexible time of dosing, Device issue, other
Reason(s) for discontinuing insulin degludec | At time of discontinuing insulin degludec (0 to 6 months)
  Reasons for discontinuing insulin degludec (if applicable and available) will be classified as: Injection site reaction, Insufficient efficacy, Hypoglycaemia (severe / non-severe / nocturnal), Weight gain, Cost, Device issue, Other

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (26):
- Canada (26):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Shubenacadie, Nova Scotia
  - Novo Nordisk Investigational Site, Sydney, Nova Scotia
  - Novo Nordisk Investigational Site, Ajax, Ontario
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Guelph, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Markham, Ontario
  - Novo Nordisk Investigational Site, Nepean, Ontario
  - Novo Nordisk Investigational Site, Oakville, Ontario
  - Novo Nordisk Investigational Site, Orillia, Ontario
  - Novo Nordisk Investigational Site, Scarborough Village, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Tecumseh, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Gatineau, Quebec
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Pierrefonds, Quebec
  - Novo Nordisk Investigational Site, Terrebonne, Quebec

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Harris SB, Ajala O, Bari B, Liutkus J, Hahn J, Martyn O, Zwicker D. Evaluating the Effectiveness of Switching to Insulin Degludec from Other Basal Insulins in a Real-World Canadian Population with Type 1 or Type 2 Diabetes: The CAN-TREAT Study. Diabetes Ther. 2021 Jun;12(6):1689-1702. doi: 10.1007/s13300-021-01063-5. Epub 2021 May 1. PMID 33932223